CLINICAL TRIAL: NCT03726242
Title: Study of Local Physiological Effects Following Intradermal and Intramuscular Injection of Levcromacalim
Brief Title: Peripheral Nociceptive Effects of Levcromakalim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, PhD student, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Levcromakalim local injection
Record Dates: First submitted 2018-10-22; First posted 2018-10-31 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Pain; Levcromakalim
MeSH Terms: conditions — Pain | interventions — Cromakalim; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel, randomized placebo controlled and crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim (Active Comparator): To investigate the role of levcromakalim compared with placebo after intradermal and intramuscular injection.
  To give 0,05 ml intradermal and 0.2 intramuscular of 150 ug/ml levcromakalim after baseline time 0.
  Interventions: Drug: Levcromakalim; Drug: Saline
- Saline (Placebo Comparator): To investigate the role of levcromakalim compared with placebo after intradermal and intramuscular injection.
  To give 0,05 ml intradermal and 0.2 intramuscular of saline after baseline time 0.
  Interventions: Drug: Levcromakalim; Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — To investigate the role of levcromakalim compared with placebo after intradermal and intramuscular injection.
Drug: Saline — To investigate the role of levcromakalim compared with placebo after intradermal and intramuscular injection.

SUMMARY:
Intradermal and intramuscular injection of levcromacalim and placebo (sterile saline) on the forehead and forearm of healthy subjects and the following will be investigated:

1. Prevalence and intensity of pain
2. Prevalence and intensity of itching
3. Occurrence and intensity of local redness and swelling
4. Occurrence and intensity of local changes in skin temperature and blood flow

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers of both sexes.
2. 18-60 years.
3. 50-100 kg.
4. Women of childbearing potential must use adequate contraception.

Exclusion Criteria:

1. A history of serious somatic disease
2. Migraine or any other type of headache (except episodic tension-type headache less than once a month)
3. Daily intake of any medication except contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Occurrence and change of pain from baseline | Before and after injection of levcromakalim compared with before and after injection of saline. Time of measurements is baseline, 5 min, 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min and 45 min after the injection
  Occurrence and intensity of pain after levcromakalim injektion compared to placebo. To measure pain numerical rating scale (NRS) 0-10 will be used.
  The outcome measure is pain and the unit that will be used to measure the pain is NRS.
Occurrence and change of Itching from baseline | Before and after injection of levcromakalim compared with before and after injection of saline. Time of measurements is baseline, 5 min, 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min and 45 min after the injection
  Occurrence and intensity of Itching after levcromakalim injektion compared to placebo. To measure itching numerical rating scale (NRS) 0-10 will be used.
  The outcome measure is itching and the unit that will be used to measure the itching is NRS.

SECONDARY OUTCOMES:
Occurrence and change of redness from baseline | Before and after injection of levcromakalim compared with before and after injection of saline. Time of measurements is baseline, 5 min, 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min and 45 min after the injection.
  Occurrence and change of redness after levcromakalim injektion compared to placebo. The areal of the redness will be measured.
  The outcome measure is redness and the unit that will be used to measure the redness is areal cm^2.
Occurrence and change of swelling from baseline | Before and after injection of levcromakalim compared with before and after injection of saline. Time of measurements is baseline, 5 min, 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min and 45 min after the injection.
  Occurrence and change of swelling after levcromakalim injektion compared to placebo. The areal of the swelling will be measured.
  The outcome measure is swelling and the unit that will be used to measure the swelling is areal cm^2.
Change of blood flow from baseline | Before and after injection of levcromakalim compared with before and after injection of saline. Time of measurements is baseline, 5 min, 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min and 45 min after the injection.
  Change of blodflow after levcromakalim injektion compared to placebo. The intensity of the blodd flow will be measured by laser speckle The outcome measure is change of blood flow and the laser speckle will be used to measure the blood flow.
Change of skin temperature from baseline | Before and after injection of levcromakalim compared with before and after injection of saline. Time of measurements is baseline, 5 min, 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min and 45 min after the injection.
  Change of skin temperature after levcromakalim injektion compared to placebo. The temperature will be measured by thermovision camera.
  The outcome measure is the change of skin temperature and the thermovision camera will be used to measure skin temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish headache center, Glostrup Municipality, Copenhagen, Denmark